CLINICAL TRIAL: NCT05488808
Title: Deep Repetitive Transcranial Magnetic Stimulation for Peripheral Neuropathic Pain. A Randomized Double-blind Sham-controlled Study.
Brief Title: Treatment of Peripheral Neuropathic Pain
Acronym: BrainStim
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Oslo University Hospital (Other)
Responsible Party: Principal Investigator, Nadine Farnes, Ph.D. student, Oslo University Hospital
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 428116
Record Dates: First submitted 2022-08-03; First posted 2022-08-05 (Actual); Last update posted 2023-11-27 (Actual); Status verified 2023-11

CONDITIONS: Neuropathic Pain
Keywords: Repetitive Transcranial Magnetic Stimulation
MeSH Terms: conditions — Neuralgia | interventions — Transcranial Magnetic Stimulation

STUDY DESIGN:
Intervention Model Description: Patients undergo stimulation with deep rTMS in a double blinded randomised controlled trial (RCT) with a 2 x 2 cross-over design, receiving both active and placebo stimulation. Patients are randomly assigned in a 1:1 ration to one of two counterbalanced arms: either they first receive active rTMS and then sham rTMS after a 9 week washout period, or the first receive sham rTMS and then active rTMS after 9 weeks of washout.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Blinding is achieved by inserting a card into the rTMS stimulator which determines whether the patient receives active or sham stimulation, making both participant and investigator blind towards group allocation. Care providers are also blinded to treatment allocation. Main efficacy analyses will be performed blinded without identification of participants and group allocation.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active and then sham rTMS (Active Comparator): Deep rTMS is delivered with the Brainsway H7-coil (Brainsway, Jerusalem, Israel) applied via a helmet placed on the head targeting the primary motor cortex of the arm.
  Interventions: Device: repetitive Transcranial Magnetic Stimulation
- Sham and the active rTMS (Sham Comparator): Sham stimulation is delivered with a sham coil placed in the helmet encasing the active rTMS coil. Sham rTMS sessions will use exactly the same parameters of stimulation as active rTMS.
  Interventions: Device: repetitive Transcranial Magnetic Stimulation

INTERVENTIONS:
Device: repetitive Transcranial Magnetic Stimulation — Deep rTMS is delivered with the Brainsway H7-coil (Brainsway, Jerusalem, Israel) applied via a helmet placed on the head targeting the primary motor cortex of the leg.

SUMMARY:
Peripheral neuropathic pain is a disabling chronic pain condition that is difficult to treat. Repetitive transcranial magnetic stimulation (rTMS) to the motor cortex is a treatment method with growing evidence in its ability to alleviate neuropathic pain. This also applies to new deep rTMS coils which permits stimulation of larger cortical areas and with deeper penetration. The aim of this study is to investigate the analgesic efficacy of 5 days of deep rTMS compared to sham stimulation. We will also assess effects of deep rTMS on sleep, psychological fatctors, everyday functioning, and executive functioning.

ELIGIBILITY:
Inclusion Criteria:

* 18-80 years of age
* Peripheral neuropathic pain related to postherpetic neuralgia, peripheral nerve injury, limb amputation, polyneuropathy or radiculopathy, fulfilling the criteria for probable or definite neuropathic pain (Finnerup et al. 2016)
* Usual pain intensity at least 4/10 over the past 24 hrs using the numerical scale of the BPI at screening
* Daily pain
* Pain for at least 3 months
* Stable pharmacological treatment for pain or no pharmaceutical treatment at least 1 month prior to inclusion participation
* Ability to follow throughout the whole duration of the study

Exclusion Criteria:

atients with phantom limb pain after limb amputation

* Any clinically significant or unstable medical or psychiatric disorder
* Subjects protected by law (guardianship or tutelage measure)
* History of or current substance abuse (alcohol, drugs)
* Pending litigation
* Contraindication to rTMS (past severe head trauma, history of epilepsy or ongoing epilepsy, active cerebral tumour, past neurosurgical intervention, intracranial hypertension, implanted devices not compatible such as cardiac pacemaker and neurostimulator, cochlear implants, pregnancy or lactation. All women of childbearing age will be required to have negative pregnancy test at inclusion and to be using contraception)
* Pain conditions more severe than peripheral neuropathic pain
* Inability to understand the protocol or to fill out the forms
* Other ongoing research protocol or recent past protocol within one month before the inclusion

Ages: 18 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 17 (Actual)
Dates: Start 2022-02-01 (Actual); Primary Completion 2023-11-24 (Actual); Study Completion 2023-11-24 (Actual)

PRIMARY OUTCOMES:
Usual pain intensity over the past 24 hours | Analgesic efficacy of active and sham treatment is measured as the change in pain intensity scores between baseline values (one week before treatment) and 1 week after the last stimulation. Measurement ends 3 weeks after last stimulation]
  Measured every day in a diary at the same hour (end of the day) on an 11-point NRS (0 = no pain, 10 = worst pain intensity imaginable of the current pain condition)

SECONDARY OUTCOMES:
Usual pain intensity over the past 24 hours | Analgesic efficacy of active and sham treatment is measured as the change in pain intensity scores between baseline values and 3 weeks after the last stimulation
  Measured every day in a diary at the same hour on an 11-point NRS (0 = no pain, 10 = worst pain intensity imaginable of the current pain condition)
Pain intensity over the last 24 hours | Baseline, 1 week and 3 weeks after the end of each stimulation period
  Maximum and minimum pain intensity hours, rated from 0 (no pain) to 10 (pain as bad as you can imagine)
Pain unpleasantness during the last 24 hours | Baseline, 1 week and 3 weeks after the end of each stimulation period
  Maximum, minimum, and usual pain unpleasantness, rated from 0 (no pain/unpleasantness) to 10 (unpleasantness as bad as you can imagine)
Intensity of dynamic mechanical allodynia | Baseline, 1 week and 3 weeks after the end of each stimulation period
  Dynamic mechanical allodynia is assessed using a brush (SOMEDIC). The outcome is the mean pain intensity of 3 brush strokes within 2 seconds intervals. The length of the brush stroke is 3 cm, measured on an 11-point NRS (0 = no pain, 10 = worst pain intensity imaginable), disregarding the spontaneous ongoing pain.
Intensity of static mechanical allodynia | Baseline, 1 week and 3 weeks after the end of each stimulation period
  Static mechanical allodynia is measured with a stimulus lightly indenting the skin for 10 seconds. The outcome is the mean pain intensity of three presses, measured on an 11-point NRS (0 = no pain, 10 = worst pain intensity imaginable), disregarding the spontaneous ongoing pain.
Proportion of responders | Baseline,1 week and 3 weeks after the end of each stimulation period]
  Proportion of responders with at least 30% and 50% usual pain intensity reduction compared to prestimulation values allowing to calculate Numbers Needed to Treat for 30 % and 50 % pain relief.
Percentage pain intensity reduction | Baseline,1 week and 3 weeks after the end of each stimulation period
  Percentage pain intensity reduction on an 11-point NRS (0 %= no pain reduction; 100% complete pain reduction)
Hospital Anxiety and Depression Scale | Baseline,1 week and 3 weeks after the end of each stimulation period
  The Hospital Anxiety and Depression Scale includes 14 items scored as anxiety and depression scores, 7 items assessing depression and 7 anxiety
Pain Catastrophizing Scale | Baseline,1 week and 3 weeks after the end of each stimulation period
  Consists of 13 items describing the occurrence of thoughts and feelings that individuals may experience when in pain rated from 0 (not at all) to 4 (all the time)
Patient Global Impression of Change | Baseline,1 week and 3 weeks after the end of each stimulation period
  Consists of 7 items to evaluate the subjective improvement or deterioration (from very much improved to very much deteriorated)
Insomnia Severity Index | Baseline,1 week and 3 weeks after the end of each stimulation period
  Consists of self-rated questions which maps sleep difficulties specific to insomnia on a 5 point Likert scale
Patient-Specific Functional Scale | Baseline,1 week and 3 weeks after the end of each stimulation period
  The Patient-Specific Functional Scale is a numeric rating scale that measures individually chosen functions that are inhibited by the pain. Patients rate from 0 (unable to perform activity) to 10 (able to perform activity)
Executive functioning using the CANTAB battery | Baseline,1 week and 3 weeks after the end of each stimulation period
  Composite score and individual analyses of the paired associates learning test, stop signal task, spatial working memory test and the multitasking test weeks after the end of each stimulation period
Side-effects | Immediately after the first rTMS session for both stimulation periods and 1 week and 3 weeks after each stimulation period
  Side effects using a specific side effects questionnaire specifically designed for assessment of safety in rTMS studies
Blinding | 3 weeks after the end of each stimulation period
  Blinding questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Audun Stubhaug, MD, PhD, Study Director — OUS
Locations (1):
- Department of Pain Management and Research, Oslo University Hospital and Faculty of Medicine, University of Oslo,, Oslo, Norway

IPD SHARING:
Plan to Share IPD: No
Deidentified individual participant data collected during the trial will be available to other researchers who provide a methodologically sound proposal, and who adhere to institutional guidelines.

REFERENCES:
- [Background] Finnerup NB, Haroutounian S, Kamerman P, Baron R, Bennett DLH, Bouhassira D, Cruccu G, Freeman R, Hansson P, Nurmikko T, Raja SN, Rice ASC, Serra J, Smith BH, Treede RD, Jensen TS. Neuropathic pain: an updated grading system for research and clinical practice. Pain. 2016 Aug;157(8):1599-1606. doi: 10.1097/j.pain.0000000000000492. PMID 27115670
- [Derived] Farnes N, Stubhaug A, Hansson P, Vambheim SM. H-Coil Repetitive Transcranial Magnetic Stimulation Relieves Pain and Symptoms of Anxiety and Depression in Patients With Chronic Peripheral Neuropathic Pain: A Randomized Sham-Controlled Crossover Study. Neuromodulation. 2024 Dec;27(8):1372-1382. doi: 10.1016/j.neurom.2024.09.002. Epub 2024 Nov 2. PMID 39488777
- [Derived] Farnes N, Jacobsen HB, Stubhaug A, Vambheim SM. H-coil repetitive transcranial magnetic stimulation does not improve executive function in patients with chronic peripheral neuropathic pain: a randomized sham-controlled crossover study. Front Psychiatry. 2024 Jul 17;15:1401008. doi: 10.3389/fpsyt.2024.1401008. eCollection 2024. PMID 39086728